CLINICAL TRIAL: NCT02562547
Title: Evaluation of the Hem-Avert® Perianal Stabilizer Into Routine Clinical Practice
Status: Completed | Type: Observational
Sponsor: Desert Perinatal Associates (Other)
Responsible Party: Sponsor
Other Study IDs: DH-SR-S-01
Record Dates: First submitted 2015-09-11; First posted 2015-09-29 (Estimated); Last update posted 2015-09-29 (Estimated); Status verified 2015-09

CONDITIONS: Cesarean Section Rate

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- All Vaginal Births: The application of the Hem-Avert Perianal Stabilizer
  Interventions: Device: Hem-Avert Perianal Stabilizer

INTERVENTIONS:
Device: Hem-Avert Perianal Stabilizer — The HEM-AVERT® Perianal Stabilizer is an FDA approved Class II device in accordance with FDA regulations 21 CFR 801.109. The HEM-AVERT® Perianal Stabilizer is a non-invasive device used to help provide continuous pressure to the perianal region as a means to help provide support during the labor process.

SUMMARY:
This is a retrospective data-only study following the phased introduction of the HEM-AVERT® Perianal Stabilizer into routine clinical practice. The investigators aim to capitalize on the introduction of the HEM-AVERT® Perianal Stabilizer into routine clinical practice in labor and delivery settings in the hospital of Dignity Health - St. Rose, Siena Campus and to determine whether the HEM-AVERT® Perianal Stabilizer reduces the frequency of Cesarean Section during labor and delivery.

DETAILED DESCRIPTION:
The on label device in this study is the HEM-AVERT® Perianal Stabilizer manufactured by Stetrix, Inc. This study is being sponsored by Dignity Health and falls within the guidelines set forth by the Food and Drug Administration in 21 CFR Section 812.2 as a non-significant risk study. The HEM-AVERT® Perianal Stabilizer is a Class II device in accordance with FDA regulation 21 CFR 801.109. Retrospective data will be collected in this study on the reduction of c-section rates and duration of second stage of labor. These data may be used to support an application to the FDA for a new indication of reducing c-sections. It is also possible the second stage labor data may also be used in support of expanded labeling.

ELIGIBILITY:
Inclusion Criteria:

* Vaginal Births

Exclusion Criteria:

* Anticipated non-vaginal birth

Sex: Female | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: Participants will be all women who present for vaginal delivery at Dignity Health - St. Rose, Siena Campus during the 3 month study period. The main focus of this study is to see whether the Hem-Avert® reduces Cesarean delivery among women undergoing labor and delivery. To be included in this study, by definition, the participant must be a pregnant woman.
Sampling Method: Probability Sample
Enrollment: 799 (Actual)
Dates: Start 2015-04; Primary Completion 2015-06 (Actual); Study Completion 2015-09 (Actual)

PRIMARY OUTCOMES:
Cesarean Conversion Rate | 90 Days
  Cesarean Conversion Rate

SECONDARY OUTCOMES:
Second stage labor times | 90 Days
  Comparing second stage labor times
Lacerations | 90 Days
  Comparing lacerations

CONTACTS AND LOCATIONS:
Overall Officials: Craig Weiner, M.D., Study Chair — Dignity Health

REFERENCES:
- [Background] Abramowitz L, Sobhani I, Benifla JL, Vuagnat A, Darai E, Mignon M, Madelenat P. Anal fissure and thrombosed external hemorrhoids before and after delivery. Dis Colon Rectum. 2002 May;45(5):650-5. doi: 10.1007/s10350-004-6262-5. PMID 12004215
- [Background] Gjerdingen DK, Froberg DG, Chaloner KM, McGovern PM. Changes in women's physical health during the first postpartum year. Arch Fam Med. 1993 Mar;2(3):277-83. doi: 10.1001/archfami.2.3.277. PMID 8252148
- [Background] Cheng CY, Li Q. Integrative review of research on general health status and prevalence of common physical health conditions of women after childbirth. Womens Health Issues. 2008 Jul-Aug;18(4):267-80. doi: 10.1016/j.whi.2008.02.004. Epub 2008 May 12. PMID 18468922
- [Background] Burns DA. Effectiveness of a novel device in the reduction of cesarean deliveries. ISRN Obstet Gynecol. 2013 Sep 1;2013:173278. doi: 10.1155/2013/173278. eCollection 2013. PMID 24078876